CLINICAL TRIAL: NCT02609126
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Trial Evaluating the Pharmacokinetics, Safety and Preliminary Efficacy of EP-104IAR (Long-Acting Fluticasone Propionate) in Patients With Osteoarthritis of the Knee
Brief Title: Safety Study of a Long-Acting Injectable Steroid to Treat Knee Osteoarthritis
Acronym: STEPUP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eupraxia Pharmaceuticals Inc. (Industry)
Collaborators: Syreon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-104IAR-101
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EP-104IAR (Experimental): 15mg EP-104IAR in 4 mL carrier fluid
  Interventions: Drug: EP-104IAR
- Vehicle (Placebo Comparator): 4 mL carrier fluid
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: EP-104IAR — Single, ultrasound-guided injection of EP-104IAR into the knee
  Arms: EP-104IAR
Drug: Vehicle — Single, ultrasound-guided injection of vehicle placebo into the knee
  Arms: Vehicle

SUMMARY:
The main purpose of this study is to understand the pharmacokinetics of EP-104IAR and to determine whether it is safe to use in patients with osteoarthritis (OA) of the knee. The study will also provide some preliminary insights into whether the experimental treatment reduces pain in the knee.

Osteoarthritis is the most common joint disease, affecting over 20 million people in the US alone. Currently, pain treatments that are injected directly into the knee often work for only a short time and may also have side effects within the rest of the body. The experimental treatment is a steroid that is in the same family of drugs as the most common current injectable treatments for knee osteoarthritis. For this study, the drug is coated with a polymer intended to prolong the time it stays inside the knee and lessen potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* OA of Index Knee
* Kellgren Lawrence Grade 2 or 3
* Patient-reported pain (PtPain) of Index Knee ≥4 but ≤9
* PtPain of non-Index Knee <6
* BMI ≦ 40 kg/m2

Exclusion Criteria:

* Intra-articular joint injection in the Index Knee within the past 8 weeks for glucocorticoids and 6 months for hyaluronic acid
* Insulin-dependent diabetes
* Active infection
* Pregnant or breast feeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of fluticasone propionate | Up to 42 weeks
Fluticasone propionate concentrations in synovial fluid | Up to 30 weeks
Area under the plasma concentration versus time curve (AUC) of fluticasone propionate | 12 weeks
Incidence of treatment-emergent adverse events | Up to 42 weeks
Change from baseline in clinical laboratory parameters: hematology, chemistry (including cortisol) and urinalysis | Up to 42 weeks

SECONDARY OUTCOMES:
Time to baseline pain in patient-reported Pain Numerical Rating Scale for Index knee | Weekly up to 42 weeks
Change from baseline in patient-reported Pain Numerical Rating Scale for Index knee | Weekly up to 42 weeks
Change from baseline in patient-reported Global Assessment of Arthritis | Up to 42 weeks
Change from baseline in patient-reported Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Up to 42 weeks
Change from baseline in patient-reported Short Form - 36 quality of life scores | Up to 42 weeks
Change from baseline in Physician's Global Assessment of Arthritis | Up to 42 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Helliwell, MD FRCPC, Study Director — Eupraxia Pharmaceuticals
Locations (3):
- Canada (3):
  - Rebalance MD, Victoria, British Columbia
  - Centre for Studies in Family Medicine, London, Ontario
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario

IPD SHARING:
Plan to Share IPD: Undecided